CLINICAL TRIAL: NCT01026571
Title: Identification of Genetic Causes of Bicuspid Aortic Valve Disease
Acronym: BAV Genetics
Status: Active, not recruiting | Type: Observational
Sponsor: Boston University (Other)
Collaborators: Massachusetts General Hospital (Other); Brigham and Women's Hospital (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Other Study IDs: H-39900; 1R21HL150373-01 (NIH)
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Bicuspid Aortic Valve
Keywords: Bicuspid aortic valve
MeSH Terms: conditions — Bicuspid Aortic Valve Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Collection of salivary DNA
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Bicuspid aortic valve: Collection of patients who are known to have bicuspid aortic valve disease, diagnosed by prior cardiac imaging
- Relative: Collection of patients who are a relative to a patient known to have bicuspid aortic valve disease, diagnosed by prior cardiac imaging

SUMMARY:
BAVgenetics is a partnership between Investigators at Boston University, Brigham and Women's Hospital, and Massachusetts General Hospital dedicated to discovering the genetic causes of bicuspid aortic valve disease and associated aortic disease.

DETAILED DESCRIPTION:
The Investigators at BAVgenetics are dedicated to discovering the mechanisms of bicuspid aortic valve disease and why individual genetics seem to play such an important role in generation of this disease.

If you have, or have had, a bicuspid aortic valve, we seek your help in this effort by volunteering to donate DNA to the BAV Registry, so that this disease can be better understood and therapies for it can be developed.

The BAV Registry is comprised of patients who have donated DNA collected from saliva (spit) and have provided us with personal health information that tells us about their bicuspid aortic valve.

Individuals in the Registry have signed the consent form, filled out the medical history questionnaire and the authorization form, and provided DNA via our saliva sample kits.

We will send you the requisite forms so that you receive the most up-to-date information about the study as older forms may be outdated. We also need paper copies of the forms; therefore, we send all the forms via ground mail along with a pre-paid return envelope for your convenience.

ELIGIBILITY:
Inclusion Criteria:

* Any adult patient ≥ 14 years of age may be recruited regardless of gender, ethnicity or racial group.
* Patients with a diagnosis of bicuspid aortic valve will be enrolled.
* Patients who have had their bicuspid aortic valve previously replaced will also be enrolled.
* Relatives of patients with a diagnosis of bicuspid aortic valve are also welcomed to be enrolled regardless if they have BAV or not, as it is helpful to examine the DNA of first degree relatives.

Exclusion Criteria:

* Non-English speaking

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The investigators wish to identify genetic variation that is associated with BAV in Americans.
  Patients with a diagnosis of bicuspid aortic valve will be enrolled. Patients who have had their bicuspid aortic valve previously replaced will also be enrolled. Relatives of patients with a diagnosis of bicuspid aortic valve are also welcomed to be enrolled regardless if they have BAV or not, as it is helpful to examine the DNA of first degree relatives.
Sampling Method: Non-Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2009-12 (Actual); Primary Completion 2029-12 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Identification of genetic variants associated with the occurrence of bicuspid aortic valve disease | 20 years

CONTACTS AND LOCATIONS:
Overall Officials: Simon C Body, MD MPH, Principal Investigator — Boston University, Anesthesiology Department
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States